CLINICAL TRIAL: NCT07083583
Title: Impact of IV Iron on Bleeding Symptoms in Iron Deficient Patients With Inherited Bleeding Disorders: a Single-arm Prospective Observational Study
Brief Title: Impact of IV Iron on Bleeding Symptoms in Iron Deficient Patients With Inherited Bleeding Disorders
Acronym: IRON-BD
Status: Recruiting | Type: Observational
Sponsor: Nicoletta C Machin (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Nicoletta C Machin, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: STUDY25020144
Record Dates: First submitted 2025-06-30; First posted 2025-07-24 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Bleeding Disorders; Iron; Platelet; Bleeding
Keywords: Iron deficiency; bleeding disorder; platelet function
MeSH Terms: conditions — Hemostatic Disorders; Hemorrhage; Iron Deficiencies | interventions — ferryl iron; Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Iron Deficient patients with underlying bleeding disorders: Subjects ≥15 years old with a history of an inherited bleeding disorder (including von Willebrand disease, platelet disorders, factor deficiencies, or bleeding disorder of unknown cause) and ferritin <50 ng/mL identified during routine clinic evaluation.
  Interventions: Drug: IV Iron (standard of care)

INTERVENTIONS:
Drug: IV Iron (standard of care) — Participants will receive IV iron therapy as part of standard management for iron deficiency

SUMMARY:
This is a prospective, single-arm, single-center observational study evaluating the impact of intravenous (IV) iron replacement in patients with inherited bleeding disorders and iron deficiency (ferritin <50ng/dL). Subjects will undergo baseline bleeding assessments, quality-of-life measures, and laboratory tests before receiving standard-of-care IV iron. Follow-up blood work and questionnaires will be conducted post-replacement to assess for changes

DETAILED DESCRIPTION:
Iron deficiency is one of the most prevalent nutritional deficiencies globally. In particular, patients with an inherited bleeding disorder are at increased risk of iron deficiency/ iron deficiency anemia given the propensity of this patient population to bleed. The impact of iron deficiency on hemoglobin synthesis is well established as it remains the leading cause of anemia worldwide, especially among menstruating women. Studies have shown a prevalence of iron deficiency as high as 93% in Hemophilia B Carriers , and iron deficiency anemia in 75% of females with von Willebrand Disease. However, platelets are also affected by iron deficiency. The effect of iron deficiency, as described in the past, is primarily seen in platelet production, where iron deficiency anemia (IDA) leads to increased platelet production or thrombocytosis. This is achieved through increased megakaryopoietic differentiation. Nonetheless, little is known about the effect of iron deficiency on platelet function and the mechanism by which it happens. In addition to that, it is unknown whether iron deficiency in patient with an underlying bleeding disorder could mitigate worsening bleeding symptoms.

Studies in mice have demonstrated that platelet function was suppressed in iron-deficient mice, with evidence of iron-dependent platelet activation promoted through calcium mobilization and αIIbβ3 activation. A recent study in women with IDA demonstrated that iron levels may affect platelet function. Flow cytometry showed that women with IDA have quiescent platelets circulating in a degranulated state, which might be refractory to hemostatic activation. That same study showed that iron repletion decreased P-selectin levels and enhanced degranulation of quiescent platelets when exposed to CRP-XL or ADP. That translated into increased adhesion to collagen. A study done in children, adolescents, and young adults highlighted that mean PFA-100 closure times were significantly longer in patients with IDA, with reduced Platelet aggregation with ADP, epinephrine, and ristocetin. That same study showed that treatment with Iron improved platelet aggregation tests and significantly decreased PFA-100.

The clinical relationship between bleeding, platelet function, and iron deficiency remains poorly understood. It is hypothesized that patients with iron deficiency may experience increased bleeding, with anecdotal evidence suggesting that bleeding improves as iron levels are restored. This effect is believed to be mediated by alterations in platelet function. However, the specific cellular and molecular mechanisms underlying platelet hyporesponsiveness in iron deficiency are poorly elucidated. This would particularly impact patients with an underlying inherited bleeding disorder who are at an increased risk of blood loss.

This study addresses the critical gap in understanding the bleeding phenotype in iron-deficient patients with inherited bleeding disorders. To date, no studies have comprehensively evaluated this relationship. The investigator proposes a prospective study to assess bleeding phenotypes through validated bleeding assessment scores and quality of life metrics, pre and post IV iron replacement. Additionally, the investigator will analyze platelet samples pre- and post-treatment to investigate the impact of iron replenishment on platelet function and hemostatic parameters. These findings will provide valuable insights into the interplay between iron deficiency, platelet function, and bleeding severity, advancing our understanding and management of this unique patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females > 15 years of age
2. Diagnosed with an Inherited Bleeding Disorder (Von Willebrand disease, platelet disorders, factor deficiencies, or bleeding disorder of unknown cause)
3. Evidence of Iron Deficiency (Ferritin < 50 ng/mL)
4. Receiving IV iron at Hemophilia Center of Western Pennsylvania
5. Willingness to have blood drawn
6. Willing to return to clinic 3 months post infusion for final blood draw, bleeding and quality of life assessments.

Exclusion Criteria:

1. Previous thrombosis, VTE History.
2. Platelet count < 100,000 * 109/L
3. Concomitant use of antiplatelet drugs, anticoagulants, aspirin, NSAIDs.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient in the outpatient setting with a bleeding disorder and Iron Deficiency planned for IV Iron as per Standard of care followed at the Hemophilia Center of Western Pennsylvania
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in bleeding assessment (ISTH-BAT score) | Baseline to 3 months post-IV iron replacement
  Change in bleeding severity 3 months after IV iron replacement, assessed using the ISTH-BAT (International Society on Thrombosis and Haemostasis Bleeding Assessment Tool).
  ISTH-BAT: Score range 0-56; higher scores indicate greater bleeding severity.
  Safety Issue:
  No
Change in Menstrual Blood Loss (PBAC Score) | Baseline to 3 months post-IV iron replacement
  Change in menstrual bleeding 3 months after IV iron replacement, measured using the Pictorial Blood Loss Assessment Chart (PBAC). Assessed only in menstruating female participants.
  PBAC: Score <100 indicates normal menstrual blood loss; scores >100 suggest heavy menstrual bleeding.
Change in Epistaxis Severity Score (ESS) | Baseline to 3 months post-IV iron replacement
  Change in epistaxis severity from baseline to 3 months post-IV iron replacement, measured using the Epistaxis Severity Score (ESS), a validated clinical tool for quantifying frequency, duration, and impact of nosebleeds.
  Score Range: 0 to 10
  Scoring Interpretation: Higher scores indicate more severe or frequent nosebleeds. A reduction in score reflects clinical improvement.

SECONDARY OUTCOMES:
Change in Fatigue (FACIT-F Score) | Baseline to 3 months post-IV iron replacement
  Change in fatigue levels from baseline to 3 months after IV iron replacement, as measured by the Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-F).
  Score Range: 0 to 160
  Scoring Interpretation: Lower scores indicate greater fatigue; higher scores indicate improved energy and well-being.
Change in Physical Functioning (SF-36) | Baseline to 3 months
  Change in physical functioning score on the SF-36 from baseline to 3 months post-IV iron.
  Score Range: 0 to 100
  Scoring Interpretation: Higher scores indicate better physical functioning.
Change in Role Limitations Due to Physical Health (SF-36) | Baseline to 3 months
  Change in score from the Role Physical domain of the SF-36, which evaluates problems with work or daily activities due to physical health.
  Score Range: 0 to 100
  Scoring Interpretation: Higher scores reflect fewer role limitations.
Change in Role Limitations Due to Emotional Problems (SF-36) | Baseline to 3 months
  Change in the Role Emotional domain score of the SF-36, which assesses limitations in daily activities due to emotional difficulties.
  Score Range: 0 to 100
  Scoring Interpretation: Higher scores indicate better emotional role functioning.
Change in the Vitality domain of the SF-36, measuring energy levels and fatigue. | Baseline to 3 months
  Change in the Vitality domain of the SF-36, measuring energy levels and fatigue.
  Score Range: 0 to 100
  Scoring Interpretation: Higher scores indicate greater energy and less fatigue.
Change in Social Functioning (SF-36) | Baseline to 3 months
  Change in the Social Functioning domain score, reflecting the extent to which physical or emotional health interferes with normal social activities.
  Score Range: 0 to 100
  Scoring Interpretation: Higher scores indicate better social functioning.
Change in Pain Score (SF-36) | Baseline to 3 months
  Change in the Bodily Pain domain of the SF-36, evaluating intensity of pain and its effect on daily activities.
  Score Range: 0 to 100
  Scoring Interpretation: Higher scores indicate less pain and better pain management.
Change in Emotional Well-Being (SF-36) | Baseline to 3 months
  Change in the Mental Health domain score of the SF-36, assessing psychological well-being, mood, and anxiety.
  Score Range: 0 to 100
  Scoring Interpretation: Higher scores indicate better emotional well-being.
Change in General Health Perception (SF-36) | Baseline to 3 months
  Change in the General Health domain score of the SF-36, which assesses overall health perceptions.
  Score Range: 0 to 100
  Scoring Interpretation: Higher scores reflect better perceived general health.

OTHER OUTCOMES:
Change in Mitochondrial Reactive Oxygen Species (ROS) in Platelets | Baseline to 3 months post-IV iron replacement
  Evaluate changes in mitochondrial reactive oxygen species (ROS) levels in platelet samples from baseline to 3 months post-IV iron replacement. This exploratory analysis will assess whether iron repletion alters platelet oxidative stress, potentially contributing to changes in platelet function and bleeding phenotype.
Change in Platelet Reactivity by Flow Cytometry | Baseline to 3 months post-IV iron replacement
  Evaluate changes in platelet reactivity before and after IV iron replacement, using flow cytometry to assess surface expression of activation markers (e.g., P-selectin, activated αIIbβ3 integrin) in response to standard agonists (e.g., ADP, CRP-XL). This exploratory analysis will examine whether iron repletion restores platelet responsiveness in iron-deficient individuals with inherited bleeding disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Nicoletta Machin, DO, Principal Investigator — University of Pittburgh
Locations (1):
- Hemophilia Center of Western Pennsylvania, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share individual participant data (IPD) that underlie the results reported in the publication, after de-identification. This may include demographic data, primary and secondary outcomes, and relevant covariates. Data will be made available to researchers who provide a methodologically sound proposal for use in academic, non-commercial research. Proposals should be directed to machinnc2@upmc.edu. Access will be granted following approval by our institutional review board or ethics committee and the execution of a data use agreement. Data will be available beginning 6 months after publication and will remain accessible for 5 years.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available beginning 6 months after publication and will remain accessible for 5 years.
Access Criteria: Proposals should be directed to machinnc2@upmc.edu. Access will be granted following approval by our institutional review board or ethics committee and the execution of a data use agreement.

REFERENCES:
- [Background] McLaughlin JM, Munn JE, Anderson TL, Lambing A, Tortella B, Witkop ML. Predictors of quality of life among adolescents and young adults with a bleeding disorder. Health Qual Life Outcomes. 2017 Apr 7;15(1):67. doi: 10.1186/s12955-017-0643-7. PMID 28388906
- [Background] Kassebaum NJ, Jasrasaria R, Naghavi M, Wulf SK, Johns N, Lozano R, Regan M, Weatherall D, Chou DP, Eisele TP, Flaxman SR, Pullan RL, Brooker SJ, Murray CJ. A systematic analysis of global anemia burden from 1990 to 2010. Blood. 2014 Jan 30;123(5):615-24. doi: 10.1182/blood-2013-06-508325. Epub 2013 Dec 2. PMID 24297872
- [Background] VanderMeulen H, Sholzberg M. Iron deficiency and anemia in patients with inherited bleeding disorders. Transfus Apher Sci. 2018 Dec;57(6):735-738. doi: 10.1016/j.transci.2018.10.015. Epub 2018 Nov 17. PMID 30470664
- [Background] Lu Z, Machin NC. 2024. Assessment of bleeding severity and prevalence of iron deficiency among hemophilia b carriers by factor ix activity levels. Blood. 144(Supplement 1):2586-2586.
- [Background] Chen YC, Chao TY, Cheng SN, Hu SH, Liu JY. Prevalence of von Willebrand disease in women with iron deficiency anaemia and menorrhagia in Taiwan. Haemophilia. 2008 Jul;14(4):768-74. doi: 10.1111/j.1365-2516.2008.01777.x. Epub 2008 May 17. PMID 18498402
- [Background] Park MJ, Park PW, Seo YH, Kim KH, Park SH, Jeong JH, Ahn JY. The relationship between iron parameters and platelet parameters in women with iron deficiency anemia and thrombocytosis. Platelets. 2013;24(5):348-51. doi: 10.3109/09537104.2012.699641. Epub 2012 Jun 27. PMID 22738419
- [Background] Liu S, Guo F, Zhang T, Zhu Y, Lu M, Wu X, He F, Yu R, Yan D, Ming Z, Shu D. Iron deficiency anemia and platelet dysfunction: A comprehensive analysis of the underlying mechanisms. Life Sci. 2024 Aug 15;351:122848. doi: 10.1016/j.lfs.2024.122848. Epub 2024 Jun 15. PMID 38885879
- [Background] Mokhtar GM, Ibrahim WE, Kassim NA, Ragab IA, Saad AA, Abdel Raheem HG. Alterations of platelet functions in children and adolescents with iron-deficiency anemia and response to therapy. Platelets. 2015;26(5):448-52. doi: 10.3109/09537104.2014.931570. Epub 2014 Jul 15. PMID 25026531
- [Background] Elstrott BK, Lakshmanan HHS, Melrose AR, Jordan KR, Martens KL, Yang CJ, Peterson DF, McMurry HS, Lavasseur C, Lo JO, Olson SR, DeLoughery TG, Aslan JE, Shatzel JJ. Platelet reactivity and platelet count in women with iron deficiency treated with intravenous iron. Res Pract Thromb Haemost. 2022 Mar 23;6(2):e12692. doi: 10.1002/rth2.12692. eCollection 2022 Feb. PMID 35356666
- [Background] Halimeh S, Rott H, Kappert G, Siebert M. 2013. Establishment of a reference range for the pbac-score. Blood. 122(21):4772-4772.
- [Background] Rodeghiero F, Tosetto A, Abshire T, Arnold DM, Coller B, James P, Neunert C, Lillicrap D; ISTH/SSC joint VWF and Perinatal/Pediatric Hemostasis Subcommittees Working Group. ISTH/SSC bleeding assessment tool: a standardized questionnaire and a proposal for a new bleeding score for inherited bleeding disorders. J Thromb Haemost. 2010 Sep;8(9):2063-5. doi: 10.1111/j.1538-7836.2010.03975.x. No abstract available. PMID 20626619